CLINICAL TRIAL: NCT00571584
Title: rFVIIa (NovoSeven®) for Treatment of Mild/Moderate Joint Bleeds in Haemophilia Patients With Inhibitors: A Double-blind Study of a Single High Dose Versus Standard Multiple Doses of rFVIIa
Brief Title: High Dose of Activated Recombinant Human Factor VII for Treatment of Mild/Moderate Joint Bleeds in Haemophilia Patients With Inhibitors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7HEAM-1510
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: activated recombinant human factor VII

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to evaluate the efficacy and safety of two dose schedules of activated recombinant human factor VII in treatment of joint bleeds in haemophilia patients with inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed of congenital haemophilia A or B with inhibitors to factor VIII or IX, respectively
* A history of 3 or more joint bleeds during the last 12 months

Exclusion Criteria:

* Joint bleeding within 7 days prior to trial start
* Treatment for bleeds within the last 5 days prior to trial start
* Clinically relevant coagulation disorders other than congenital haemophilia A or B

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-11; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Global treatment response of the patient by an algorithm based pain and joint mobility assessments

SECONDARY OUTCOMES:
Pain assessment
Mobility assessment
Circumference of joint
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (16):
- France (4):
  - Novo Nordisk Investigational Site, Le Kremlin-Bicêtre
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Lyon
  - Novo Nordisk Investigational Site, Paris
- Novo Nordisk Investigational Site, Budapest, Hungary
- Novo Nordisk Investigational Site, Tel Litwinsky, Israel
- Poland (3):
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
- Spain (2):
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Valencia
- Turkey (Türkiye) (2):
  - Novo Nordisk Investigational Site, Bornova-IZMIR
  - Novo Nordisk Investigational Site, Capa-ISTANBUL
- United Kingdom (3):
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Canterbury
  - Novo Nordisk Investigational Site, Sheffield

REFERENCES:
- [Result] Kavakli K, Makris M, Zulfikar B, Erhardtsen E, Abrams ZS, Kenet G; NovoSeven trial (F7HAEM-1510) investigators. Home treatment of haemarthroses using a single dose regimen of recombinant activated factor VII in patients with haemophilia and inhibitors. A multi-centre, randomised, double-blind, cross-over trial. Thromb Haemost. 2006 Apr;95(4):600-5. PMID 16601828
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com